CLINICAL TRIAL: NCT03563586
Title: Prospective Randomized Monocentric Trial of Mechanical Bowel Preparation Alone vs Mechanical Bowel Preparation Combined With Oral Antibiotics Before Colorectal Resections for Cancer
Brief Title: Mechanical Bowel Preparation With or Without Oral Antibiotics for Colorectal Cancer Surgery
Acronym: MECCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, George Theodoropoulos, Associate Professor, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 56/14-3-2018
Record Dates: First submitted 2018-06-09; First posted 2018-06-20 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Antibiotic; Bowel Cancer; Colorectal Cancer; Surgical Site Infection
Keywords: oral antibiotic; mechanical bowel preparation; colorectal cancer; surgical site infection
MeSH Terms: conditions — Intestinal Neoplasms; Colorectal Neoplasms; Surgical Wound Infection | interventions — Anti-Bacterial Agents; Cathartics

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bowel Preparation plus antibiotics (Active Comparator): Preoperative oral antibiotic therapy with rifaximin 400 mg plus metronidazole 500mg the day prior to surgery at 2:00, 3:00 and 10:00 pm, with mechanical bowel preparation (2 vials sodium phospate 45ml at 1:00 and 7:00 pm)
  Interventions: Other: Bowel Preparation plus antibiotics
- Bowel Preparation (Other): Preoperative mechanical bowel preparation (2 vials sodium phospate 45ml at 1:00 and 7:00 pm)
  Interventions: Other: Bowel Preparation

INTERVENTIONS:
Other: Bowel Preparation plus antibiotics — Preoperative oral antibiotic therapy with rifaximin 400 mg plus metronidazole 500mg the day prior to surgery at 2:00, 3:00 and 10:00 pm, with mechanical bowel preparation (2 vials sodium phospate 45ml at 1:00 and 7:00 pm)
  Arms: Bowel Preparation plus antibiotics
Other: Bowel Preparation — Mechanical Bowel Preparation (2 vials sodium phospate 45ml at 1:00 and 7:00 pm) alone Both groups will receive iv antibiotics (cefoxitin 2 gr plus metronidazole 500gr) perioperatively and discontinuation within 24 hours
  Arms: Bowel Preparation

SUMMARY:
Investigation of the role of adding oral antibiotics to preoperative mechanical bowel preparation before colorectal surgery for cancer.

DETAILED DESCRIPTION:
The aim of the study is to investigate whether the addition of oral antibiotics to Mechanical Bowel Preparation (MBP) prior to colorectal cancer surgical procedures reduce the superfical and deep surgical site (SSI) infectious complications. The study is prospective and is designed in a randomized single-blinded controlled fashion. It is taking place at one academic surgical unit of Athens Medical School, located at a tertiary referal institution. Patients scheduled to undergo an elective surgical resection for colon or rectal cancer will be allocated to either formal MBP the day before surgery or a combined MBP with administration of oral antibiotics. Exclusion criteria are the following: emergency surgery, obstructive or perforated cancer, patients intolerance to bowel preparation regimen and allergies to orally administered antibiotics.

Intervention arms: Patients will be randomised into two groups, concealed from the treating surgeon.

Group A:

Preoperative oral antibiotic therapy with rifaximin 400 mg plus metronidazole 500mg the day prior to surgery at 2:00, 3:00 and 10:00 pm, with MBP (2 vials sodium phospate 45ml at 1:00 and 7:00 pm)

Group B:

MBP (2 vials sodium phospate 45ml at 1:00 and 7:00 pm) alone Both groups will receive iv antibiotics (cefoxitin 2 gr plus metronidazole 500gr) perioperatively and discontinuation within 24 hours.

Outcome measures: The primary end point is surgical site infection (SSI), including (i) superficial wound infection, (ii) deep wound infection, and (iii) intrabdominal infection (contaminated fluid or pus collection) within 30 days of the procedure (decrease 3% in the rate) Secondary measures: Anastomotic leaks, other surgical and non-surgical compliactions, hospital length of stay, readmission rate, patients' preparation tolerance, preparation regimens side-effects, time to beginning of adjuvant treatment for colorectal cancer.

Sample Size: It is estimated that 105 patients per treatment arm are needed.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled colorectal cancer surgery

Exclusion Criteria:

* Emergency surgery
* Obstructive and perforated cancer
* Intolerance to bowel preparation regimen
* Allergies to orally administered antibiotics

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infections | 30 days
  Surgical Site Infections

SECONDARY OUTCOMES:
Anastomotic leaks | 30 days
  Anastomotic leaks
Other surgical and non-surgical compliactions | 30 days
  Other surgical and non-surgical compliactions
Hospital length of stay | 30 days
  Hospital length of stay
Readmission rate | 30 days
  Readmission rate
Patients' preparation tolerance | 30 days
  Patients' preparation tolerance
Preparation regimens side-effects | 30 days
  Preparation regimens side-effects
Time to beginning of adjuvant treatment for colorectal cancer | 60 days
  Time to beginning of adjuvant treatment for colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: George Theodoropoulos, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- NKUAthens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frountzas M, Michalopoulou V, Georgiou G, Kanata D, Matiatou M, Kimpizi D, Matthaiou G, Spiliotopoulos S, Vouros D, Toutouzas KG, Theodoropoulos GE. The Impact of Mechanical Bowel Preparation and Oral Antibiotics in Colorectal Cancer Surgery (MECCA Study): A Prospective Randomized Clinical Trial. J Clin Med. 2024 Feb 19;13(4):1162. doi: 10.3390/jcm13041162. PMID 38398474
- [Derived] Willis MA, Toews I, Soltau SL, Kalff JC, Meerpohl JJ, Vilz TO. Preoperative combined mechanical and oral antibiotic bowel preparation for preventing complications in elective colorectal surgery. Cochrane Database Syst Rev. 2023 Feb 7;2(2):CD014909. doi: 10.1002/14651858.CD014909.pub2. PMID 36748942